CLINICAL TRIAL: NCT00273429
Title: Cosopt Versus Xalatan
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pharmaceutical Research Network (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PRN 04-015
Record Dates: First submitted 2006-01-06; First posted 2006-01-09 (Estimated); Last update posted 2007-01-09 (Estimated); Status verified 2007-01

CONDITIONS: Open-Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — dorzolamide

INTERVENTIONS:
Drug: timolol maleate 0.5%
Drug: dorzolamide/timolol maleate fixed combination
Drug: latanoprost 0.005%
Drug: placebo

SUMMARY:
To compare the 24-hour efficacy and safety, measured every three hours, of the dorzolamide/timolol fixed combination given twice daily versus latanoprost and placebo each given once daily.

ELIGIBILITY:
Inclusion Criteria:

* adults with primary open-angle, pigmentary, or exfoliation glaucoma, or ocular hypertenstion
* intraocular pressure should be 22 to 30 mm Hg inclusive on timolol BID at the 08:00 H
* ETDRS visual acuity must be 1.0 or better in both eyes

Exclusion Criteria:

* any contraindications to study medications
* any anticipated change in systemic hypertensive therapy during the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-04; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: William C. Stewart, MD, Study Director — Pharmaceutical Research Network, LLC; Jay Mulaney, MD, Principal Investigator — Central Florida Eye Associates; Sriram Sonty, MD, FACS, Principal Investigator — Midwest Eye Center SC
Locations (2):
- United States (2):
  - Central Florida Eye Associates, Lakeland, Florida
  - Midwest Eye Center SC, Bourbonnais, Illinois